CLINICAL TRIAL: NCT03117127
Title: The Consumption of Whole Eggs Versus Egg Whites to Stimulate Postprandial Muscle Protein Synthesis
Brief Title: Muscle Protein Synthesis After Whole Egg vs. Egg White Consumption
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Urbana-Champaign (Other)
Responsible Party: Principal Investigator, Nicholas Burd, Assistant Professor, University of Illinois at Urbana-Champaign
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 15693
Record Dates: First submitted 2017-04-10; First posted 2017-04-17 (Actual); Last update posted 2018-05-01 (Actual); Status verified 2018-04

CONDITIONS: Hypertrophy
MeSH Terms: conditions — Hypertrophy | interventions — Resistance Training; Egg White

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Whole eggs (Active Comparator): After resistance exercise, participants will ingest whole eggs (18 g protein, 17 g fat) cooked in scrambled form.
  Interventions: Behavioral: Resistance Exercise; Other: Whole Eggs
- Egg Whites (Experimental): After resistance exercise, participants will ingest egg whites (18 g protein, 0 g fat) cooked in scrambled form.
  Interventions: Behavioral: Resistance Exercise; Other: Egg Whites

INTERVENTIONS:
Behavioral: Resistance Exercise — Participants will perform leg extension and leg press immediately prior to ingestion of whole eggs or egg whites
Other: Whole Eggs — Participants will ingestion whole eggs immediately after resistance exercise
  Arms: Whole eggs
Other: Egg Whites — Participants will ingestion whole eggs immediately after resistance exercise
  Arms: Egg Whites

SUMMARY:
In crossover trials, ten (N=10) young men (18-35 y) will receive stable isotope tracer infusions and perform a single bout of resistance exercise. Immediately after resistance exercise, participants will ingest stable isotope labeled whole eggs (18 g protein, 17 g fat) or egg whites (18 g protein, 0 g fat) cooked in scrambled form. Repeated blood and muscle biopsies will be collected to determine whole body amino acid kinetics, muscle amino acid transporters, anabolic signaling and myofibrillar protein synthesis rates during the trials.

DETAILED DESCRIPTION:
On both infusion trials, participants will report to the laboratory at 0700 h after an overnight fast. Upon arrival to the lab, a baseline breath sample will be collected for determination of 13CO2 enrichment by isotope ratio mass spectrometry. A Teflon catheter will be inserted into an antecubital vein for baseline blood sample collection (t=-210 min) and then participants will receive priming doses of NaH13CO2 (2.35 µmol·kg-1), L-[1-13C]leucine (7.6 µmol·kg-1), and L-[ring-2H5]phenylalanine (2.0 µmol·kg-1). Subsequently, a continuous intravenous infusion of L-[1-13C]leucine (0.10 µmol·kg-1·min-1) and L-[ring-2H5]phenylalanine (0.05 µmol·kg-1·min-1) will be initiated (t=-210 min) and maintained over the infusion trials. A second Teflon catheter willinserted into a heated dorsal hand vein for repeated arterialized blood sampling and remained patent by a 0.9% saline drip. Breath samples and arterialized blood samples and will be collected every 30 or 60 min during the postabsorptive- and postprandial states. In the post-absorptive state of infusion trial 1, muscle biopsies will be collected at t=-150 and -30 min of infusion to determine basal-state myofibrillar protein synthesis rates, relative skeletal muscle amino acid transporter content, and anabolic-related signaling. In the subsequent cross-over trial only 1 muscle biopsy will be collected at t=-30 for Western blot analysis and postabsorptive myofibrillar protein-bound tracer enrichment. After collection of the resting muscle biopsy at t=-30 for both trials, the participants will perform resistance exercise that consists of 4 sets of 10 repetitions at 80% of 10-RM for both leg press and leg extension exercise.

Immediately after completion of the exercise bout, participants will consume 3 whole eggs or an equivalent amount of protein from egg whites (t=0 min). Completion of the meal will mark the start of the postprandial phase (t=0 min) and additional muscle biopsies will be collected at t=120 and 300 min.

ELIGIBILITY:
Inclusion Criteria:

* Male
* Aged 18-35 years
* Healthy, active (self-reported to exercise 2 - 4 times per week)
* BMI > 18.5 and < 25 kg/m2

Exclusion Criteria:

* Smoking
* Known allergies to egg consumption
* Vegans
* Diagnosed GI tract diseases
* Arthritic conditions
* A history of neuromuscular problems
* Diagnosed cognitive impairments
* Recent (1 year) participation in amino acid tracer studies
* Predisposition to hypertrophic scarring or keloid formation
* Individuals on any medications known to affect protein metabolism (i.e. corticosteroids, non-steroidal anti-inflammatories, or prescription strength acne medications).
* High blood pressure (Systolic > 140 mm HG; Diastolic > 90 mm HG)

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Estimated)
Dates: Start 2015-07 (Actual); Primary Completion 2017-02 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
Fractional synthetic rate of myofibrillar proteins to whole egg and egg white ingestion | Postabsorptive for 3 hours, Postprandial for 5 hours
  Myofibrillar protein synthesis rates will be assessed during the postabsorptive period for 3 hr and during the 5 hr after the ingestion of the experimental beverages. This will allow us to assess the change from the postabsorptive to the postprandial period

SECONDARY OUTCOMES:
Phosphorylation of muscle anabolic signaling | Baseline and at 2 and 5 hours after protein ingestion
  Phosphorylation of anabolic signaling pathways will be assessed in the fasted state and at 2 and 5 hr after the ingestion of the whole egg and egg whites
Exogenous rate of leucine appearance after ingestion of whole eggs and egg whites. | 5 hour postprandial phase
  Dietary derived leucine availability will be measured during the 5 h postprandial phase to compare the dietary-derived leucine availability after whole egg and egg white ingestion.

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas A Burd, Ph.D., Principal Investigator — Assistant Professor
Locations (1):
- Freer Hall, Urbana, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] van Vliet S, Shy EL, Abou Sawan S, Beals JW, West DW, Skinner SK, Ulanov AV, Li Z, Paluska SA, Parsons CM, Moore DR, Burd NA. Consumption of whole eggs promotes greater stimulation of postexercise muscle protein synthesis than consumption of isonitrogenous amounts of egg whites in young men. Am J Clin Nutr. 2017 Dec;106(6):1401-1412. doi: 10.3945/ajcn.117.159855. Epub 2017 Oct 4. PMID 28978542